CLINICAL TRIAL: NCT07093086
Title: A Single-arm, Open-label Clinical Study Evaluating the Efficacy and Safety of CD20/CD19/CD22 Multi-targeted Chimeric Antigen Receptor T-cell (CAR-T) Injection in Patients With Relapsed/Refractory B-cell Lymphoma.
Brief Title: Clinical Study of Multi-targeted CAR-T Therapy in Patients With Relapsed/Refractory B-Cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U05
Record Dates: First submitted 2025-07-21; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: B-cell Lymphoma
Keywords: CAR-T; CD19; CD22; CD20
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-targeted CAR-T Therapy (Experimental): Patients will receive a regimen combining CD19/CD22 dual-targeted CAR-T cells with CD19/CD20 dual-targeted CAR-T cells; investigators may administer them sequentially according to each patient's condition.
  Interventions: Drug: Triple-targeted CAR-T Therapy

INTERVENTIONS:
Drug: Triple-targeted CAR-T Therapy — Lymphodepletion preconditioning is required prior to CAR-T cell therapy. Lymphodepletion will be performed using a regimen of cyclophosphamide (250-500 mg/m²) and fludarabine (25-30 mg/m²), each administered for 3 consecutive days.

SUMMARY:
This is a single-arm, open-label clinical study evaluating the efficacy and safety of CD20/CD19/CD22 multi-targeted chimeric antigen receptor T-cell (CAR-T) injection in patients with relapsed/refractory B-cell lymphoma.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety and efficacy of CD19/CD20/CD22 muti-target CAR-T therapy in patients with relapsed or refractory B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent obtained from the participant (or legally authorized representative) with good compliance expected throughout the study.
2. All of the following must be fulfilled:

   1. Age 2-75 years at the time of informed consent; both sexes eligible.For minors (≤18 years), consent must be provided by a parent or legal guardian; minors who are able to sign must co-sign with their guardian.
   2. Histologically confirmed B-cell lymphoma according to the NCCN Clinical Practice Guidelines in Oncology: B-Cell Lymphomas (2024 v3).
   3. Relapsed or refractory B-cell lymphoma after at least two prior lines of therapy (one standard chemo-regimen + one salvage regimen) that must have included:

      * anti-CD20 monoclonal antibody (except for subjects with documented CD20-negative tumors), and
      * an anthracycline-containing regimen.

   Subjects must additionally meet at least one of the following:

   i. Ineligible for autologous hematopoietic stem-cell transplantation (ASCT); ii. Refusal of ASCT; iii. Relapse after ASCT. d) Disease status at screening:

   • Relapse: progression after prior response (PR or CR).

   • Refractory: i. No response to last therapy (progressive disease [PD] during/after, or best response ≤SD lasting <6 months); OR ii. Relapse or progression after ASCT (biopsy-proven) including: relapse/PD ≤12 months post-ASCT, or relapse/PD after salvage therapy post-ASCT without response (SD or PD).
3. Tumor tissue (archival or fresh biopsy) positive for CD20 and/or CD19 and/or CD22 by immunohistochemistry (pathology report within 6 months preferred).
4. ≥1 measurable lesion per Lugano 2014 (Cheson) criteria.
5. ECOG performance status 0-3.
6. Adequate marrow reserve at screening:Absolute lymphocyte count (ALC) ≥0.3 × 10⁹/L; Platelets ≥30 × 10⁹/L (transfusion permitted).
7. Adequate organ function:AST ≤3×ULN (≤5×ULN if attributable to tumor infiltration); ALT ≤3×ULN (≤5×ULN if attributable to tumor infiltration); Total bilirubin ≤2×ULN (≤3×ULN with direct bilirubin ≤1.5×ULN for Gilbert's syndrome); Serum creatinine ≤1.5×ULN or creatinine clearance ≥60 mL/min (Cockcroft-Gault); Pulmonary reserve: ≤Grade 1 dyspnea and SpO₂ >91 % on room air; LVEF ≥50 % by echocardiography; INR ≤1.5×ULN and APTT ≤1.5×ULN.
8. Women of child-bearing potential must have a negative serum/urine pregnancy test within 7 days before CAR-T infusion. All participants with reproductive potential must use effective contraception from screening through at least 12 months after the last CAR-T dose.
9. Adequate venous access for leukapheresis or repeated phlebotomy, with no contraindications to leukapheresis.
10. Anticipated survival ≥3 months.

Exclusion Criteria:

1. Concurrent malignancy other than the study indication. Exceptions: carcinoma in situ or any malignancy with disease-free survival ≥3 years.
2. Use of immunosuppressive agents or systemic corticosteroids within 1 week before leukapheresis that, in the investigator's judgment, could substantially impair T-cell function.
3. Presence of any of the following:• Positive HBe-Ab and/or HBc-Ab with HBV-DNA above the lower limit of quantification;• Positive HCV-Ab with HCV-RNA above the lower limit of quantification;• Positive Treponema pallidum antibody (TP-Ab);• Positive HIV antibody.
4. Active bacterial, fungal, viral, mycoplasmal, or other infection that, in the investigator's opinion, cannot be adequately controlled.
5. Prior or current CNS disorders unrelated to lymphoma-e.g., seizure disorder, cerebral ischemia/hemorrhage, dementia, cerebellar disease, or any CNS autoimmune disease-deemed uncontrolled by the investigator.
6. Within 12 months before informed consent: percutaneous coronary intervention (angioplasty or stent placement), or NYHA Class III-IV congestive heart failure, or history of myocardial infarction, unstable angina, or other clinically significant cardiac disease judged by the investigator. QTc interval >480 ms (Fridericia correction), or left-ventricular ejection fraction <50 % by echocardiography at screening.
7. Known primary immunodeficiency.
8. History of severe immediate hypersensitivity to any study-related drug.
9. Receipt of any live vaccine within 6 weeks before screening.
10. Pregnant or breastfeeding women.
11. Active autoimmune disease requiring systemic immunosuppressive therapy.
12. Participation in any other interventional clinical trial within 30 days before signing informed consent.
13. Any condition that, in the investigator's opinion, renders the subject unsuitable for study participation.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2026-12-18 (Estimated); Study Completion 2028-12-18 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events after CAR-T cells infusion [Safety and Tolerability] | 28 days post administration of CAR-T-cells
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Objective Response Rate (ORR), as assessed by Investigators | 2 years post CAR T cell infusion
  The Objective Response Rate (ORR) is the percentage of participants who achieved a best overall response of Complete Remission (CR) or Partial Remission (PR)
Duration of response (DOR), as assessed by Investigators | 2 years post CAR T cell infusion
  Duration of response (DOR) is defined as the time from the first documented objective response to the first documented disease progression or death.
Progression-free survival (PFS), as assessed by Investigators | 2 years post CAR T cell infusion
  Progression-free survival (PFS) was defined as the time from the date of infusion to the earliest date of the first objective documentation of progressive disease (PD) or death due to any cause.
Overall survival (OS) | 2 years post CAR T cell infusion
  Overall Survival (OS) was defined as the time from the date of first infusion to the date of death due to any cause.

SECONDARY OUTCOMES:
Pharmacokinetics of CAR-T cells | 2 years post CAR T cell infusion
  Time at the maximal concentration(Tmax)
Pharmacokinetics of CAR-T cells | 2 years post CAR T cell infusion
  Area under the concentration-time curve(AUC)
Pharmacokinetics of CAR-T cells | 2 years post CAR T cell infusion
  The maximal concentration of peripheral blood (Cmax)
Pharmacodynamics of CAR-T cells | 2 years post CAR T cell infusion
  Concentration levels of CAR-T-related serum cytokines such as IL-6, IFN γ, ferritin and CRP at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Junfang Yang, Ph.D., Principal Investigator — Hebei Yanda Ludaopei Hospital
Locations (2):
- China (2):
  - Hebei Yanda Ludaopei Hospital, Hebei
  - Tongji Hospital of Tongji University, Shanghai